CLINICAL TRIAL: NCT04320693
Title: Expanded Access for IMMU-132
Status: Approved for marketing | Type: Expanded Access
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: IMMU-132
Record Dates: First submitted 2020-03-19; First posted 2020-03-25 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2020-04

CONDITIONS: Metastatic Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — sacituzumab govitecan

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: IMMU-132 — IMMU-132 will be administered as an intravenous infusion on Days 1 and 8 of 21-day treatment cycles
  Other Names: Sacituzumab Govitecan

SUMMARY:
This is an expanded access program (EAP) for eligible participants designed to provide access to IMMU-132.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult